CLINICAL TRIAL: NCT00935298
Title: Prospective Study:Clinical Trial on the Tacrolimus Dosage Range in Chinese Renal Transplant Recipients With Different Genetic Phenotypes of Drug Metabolizing Enzymes(CYP3A5)
Brief Title: Initial Dosage Range of Tacrolimus by Genotyping in Chinese Renal Transplantation
Acronym: PSIDRTG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Artillery General Hospital (Other)
Collaborators: Capital Medical University (Other); Shanghai Changzheng Hospital (Other); Pharmacology Research Institute (Other); Air Force General Hospital of the PLA (Other Government); Health Department of General Logistics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20071016; 20090403
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Tacrolimus; CYP3A5; Genotyping
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T (Experimental): The genotyping of gene CYP3A5 will be carried out in the 4-7days before renal transplantation.After transplantation, the patients will be treated by MMF, corticosteroids and tacrolimus at a dosage adapted to their genotype(CYP3A5*1/*3 and *1/*1 ,expressors; CYP3A5*3/*3 nonexpressor）.
  The objective is to determine the initial dosage Range of tacrolimus in Chinese renal transplantation patients by genotyping of the cytochrome P450 3A5
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — The genotyping of gene CYP3A5 will be carried out in the 4-7days before renal transplantation. After transplantation, the patients will be treated by MMF, corticosteroids and tacrolimus at a dosage adapted to their genotype(CYP3A5*1/*1 type and CYP3A5*1/*3 type administer 0.15mg/kg/d，CYP3A5*3/*3 type administer 0.08mg/kg/d).
  Other Names: Prograf® capsules (tacrolimus)

SUMMARY:
Acute rejection (AR) is the main complication after transplantation, which is a severe risk of chronic rejection and implant devitalization.

Tacrolimus (FK506) is an immunosuppressant used for the prevention of episodes of acute rejection. Tacrolimus is characterized by a narrow therapeutic index and important interindividual variations of its pharmacokinetic characteristics.

Tacrolimus is metabolized through the liver by the cytochrome P450 system, the cytochrome P450 3A5 (CYP 3A5) isoenzyme specifically. Polymorphisms in the CYP 3A5 gene have been associated with changes in metabolic function of the translated isoenzyme. These polymorphisms result in metabolism acceleration of tacrolimus as compared to subjects having the wild type gene, consequently leading to insufficiency of tacrolimus; it is theorized that this leads to higher risk of acute rejection. Several retrospective studies suggested an association between a genetic polymorphism of CYP3A5 and the interindividual variations of tacrolimus blood concentration. In particular, our initial study showed that adult renal transplant recipients with the CYP3A5*1/*3 and *1/*1 （expressors） genotype require higher, fixed, starting dose compared with CYP3A5*3/*3 （nonexpressor）to reach the predefined target exposure early after transplantation.

This prospective study is designed to evaluate whether genetic testing of CYP 3A5 can improve tacrolimus initiation better than usual care. This study is a prospective, multicentric, open, parallel , efficacy study. 300 receivers of a renal transplant in 8 centres will be included.

The genotyping of gene CYP3A5 will be carried out in the 4-7days before renal transplantation. After transplantation, the patients will be treated by MMF, corticosteroids and tacrolimus at a dosage adapted to their genotype(0.15mg/kg/d for CYP3A5*1/*1 type and CYP3A5*1/*3 type，0.08mg/kg/d for CYP3A5*3/*3 type).

The determination of tacrolimus blood concentration will be carried out on Day 3,5,7,14,18,21,28,35,49,63,77,90. The daily amounts of tacrolimus could be modified if necessary to reach the desired blood concentrations. The total duration of the study for a patient is 3 months after transplantation.

The objective of this study is to determine the initial dosage of tacrolimus in Chinese renal transplantation patients by genotyping of the cytochrome P450 3A5

DETAILED DESCRIPTION:
VISITS

The participation of the patient in this study will be 3 months. For this period, 9 visits are planned

•Before transplantation

Visit 1: inclusion visit(in the 4-7 days before transplantation),A blood taking will be carried out on EDTA tube for CYP 3A5 genotyping in the 4-7 days before renal transplantation.

• After transplantation

Visit 2: D3

Visit 3: D5

Visit 4: D7

Visit 5: D14

Visit 6: D21

Visit 7: M1 + - 3 days

Visit 8: M2 + - 3 days

Visit 9: M3 + - 3 days

Treatment

After transplantation, the patients will be treated by MMF, corticosteroids and tacrolimus at a dosage adapted to their genotype(CYP3A5*1/*1 type and CYP3A5*1/*3 type administer 0.15mg/kg/d，CYP3A5*3/*3 type administer 0.08mg/kg/d).

The MMF will be given according to weight in 3 months after transplantation as follows:

below 50 kilogram(kg) 0.25g bid (0.5g pre day)

50~70kg 0.50g bid (1.0g pre day)

70~90kg 0.75g bid (1.5g pre day)

Exceed 90kg 1.0g bid (2.0g pre day)

Corticosteroid therapy in decreasing amount as follows:

D0 - D15: 20 Mg

D16 - D30: 15 Mg

D30 - D45: 10 Mg

D46 - M3 5 Mg

The determination of tacrolimus blood concentration will be carried out on Day 3,5,7,14,18,21,28,35,49,63,77,90. The daily amounts of Tacrolimus could be modified if necessary to reach the desired blood concentrations. The total duration of the study for a patient is 3 months after transplantation.

If the present study is able to confirm an advantage for a genotype-driven algorithm, in terms of improved efficiency, therapeutic efficacy, especially, safety, a pharmacogenetics approach to dosing can be recommended as the basis wide quality improvement initiative that should improve patient outcomes, reduce resource use (costs of achieving safe and therapeutic immunosuppression), and reduce adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Patients of renal inadequacy , necessary to receive renal transplantation , male or female , 18 to 65 years old;
* Patients receiving a first isolated renal graft with administration of FK506;
* Patient willing to provide informed consent prior to the specimen collection procedure.

Exclusion Criteria:

* Patients who received another clinical pharmaceutical study less than 3 months before the entry in this study , and who have already completed or dropped out of this study.
* Patients with contraindications of FK506 in immunosuppressive therapy : being in pregnancy and being allergic or intolerant with FK506 or other macrolides.
* Patients suffering from severe diseases of cardiovascular system (essential hypertension), liver (anamnesis of type B hepatitis , type C hepatitis) , hemopoietic system , nervous system , and psychotics.
* Patients interfered with their blood concentrations of FK506 by administration of cytochrome P4503A4 and P4503A5 enzyme inhibitors , such as lidocaine , midazolam , nicardipine , niludipine , cortisone , itraconazole , fluconazole , ketoconazole , miconazole , clotrimazole ，Bromocriptine and so on.
* Patients having anaemia (hemoglobin lower than 7g/dl).
* Patients Diagnosed DM.
* Patients interfered with their capacity to absorb FK506 by anorexia nervosa , malabsorption syndrome or gastro-intestinal resection according to the viewpoint of the investigators.
* Patients who lacks understanding of the medicinal knowledge of tacrolimus and the risks of the study according to the viewpoint of the investigators.
* Patients with allergic constitution or a history of serious allergy.
* Patients with bad compliance according to viewpoint of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The time to obtain first target concentration of FK506 (8-13ng/ml) | 1w
  The interval time (median) after transplantation to achieve first target tacrolimus blood concentration range (7~13ng/ml) by genotype was 7 days (3 to 28) for CYP3A5*1/*3&*1/*1 patients (N=59) and 3 days (3 to 14) for CYP3A5 *3/*3 patients (N=86)
The proportion of patients reaching therapeutic concentration on Day 3 and 7 without dosage schedule adjustments | 1 w
  As compared with patients with cyp3A5*1/*3 (expression，n=59)，patients with the CYP3A5*3/*3 (nonexpression, n=86) had a decreased time to the first tacrolimus blood concentration within the therapeutic range，but had a increased proportion of patients reaching therapeutic range on Day 3-7 after tranplantration（91.8% vs. 64.4%，P = 0.021).

SECONDARY OUTCOMES:
The total number of determination of FK506 therapeutic concentration (for safety, efficiency or dose insufficiency reasons) | 3 months
  Tacrolimus blood concentration were measured 1566 times
After transplantation,the average daily tacrolimus dose, occurrence of acute rejection，delayed renal graft events | 3months
  There were one acute rejection and thirteen delayed renal allograft function events involving 14 patients, The acute rejection event occurred within the first 14 days after the initiation of tacrolimus treatment at a mean dose of 0.11 mg/kg per day and a median TBC of 4.5ng/ml (range, 3.2 to 6.2ng/ml),and this patient was heterozygous for CYP3A5*1/*3.
  Thirteen delayed renal allograft function occurred within the first 3 months including in 5 patients with CYP3A5*1/*3 genotype and in 8 patients with CYP3A5*3/*3 genotype.
Survival of the grafts at M3 | 3months
  In three months, 145 cases, 144 patients survived
Duration of the hospitalizations during the first 3 months | 3 months
  The average length of hospitalization for CYP3A5 *3/*3 and CYP3A5 *1/*3& *1/*1 patients were 38 days and 35 days, respectively (P>0.05) ,sod there was no statistically significant difference.

CONTACTS AND LOCATIONS:
Overall Officials: LIHong LIU, MD Ph.D, Study Chair — The Second Artillery Genaral Hospital
Locations (5):
- China (5):
  - Chaoyang Hospital, affiliated Hospital of Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of Air Force of Chinese PLA, Beijing, Beijing Municipality
  - The Second Artillery Gernal Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Changzheng Hospital, the Second Affiliated Hospital of the Second Military Medical University, Shanghai, Shanghai Municipality